CLINICAL TRIAL: NCT06974617
Title: Sphenopalatine Block Versus BOTOX in Management of Chronic Migraine: A Randomized Clinical Trial
Brief Title: Sphenopalatine Block Versus BOTOX in Management of Chronic Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Elsaid Abdel Fattah, Lecturer of Anesthesia, Surgical ICU and Pain Management, Faculty of Medicine, National Cancer Institute, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP2411-501-101-193
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Sphenopalatine Block; BOTOX; Chronic Migraine
MeSH Terms: interventions — Sphenopalatine Ganglion Block; Lidocaine; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sphenopalatine block group (Experimental): Patients will receive 2 ml of 2% lidocaine using a nasal applicator in each nostril.
  Interventions: Drug: Sphenopalatine block
- BOTOX group (Experimental): Patients will receive Botulinum Toxin Type A 100 units administered in a fixed dose and site paradigm.
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Sphenopalatine block — Patients will receive 2 ml of 2% lidocaine using a nasal applicator in each nostril.
  Other Names: Lidocaine
  Arms: Sphenopalatine block group
Drug: Botulinum Toxin Type A — Patients will receive Botulinum Toxin Type A 100 units administered in a fixed dose and site paradigm.
  Arms: BOTOX group

SUMMARY:
This trial compares the efficacy and safety of sphenopalatine ganglion block (SPGB) and intramuscular BOTOX injection in chronic migraine.

DETAILED DESCRIPTION:
The International Headache Society's Headache Classification Committee recognizes three broad categories of headaches: primary headaches, secondary headaches, and a third catchall category called "painful cranial neuropathies, other facial pain, and other headaches." Migraines fall into the primary headache category.

Sphenopalatine ganglion (SPG), or the pterygopalatine ganglion (PPG), is a large extracranial parasympathetic ganglion with multiple neural connections, including autonomic and motor.

The botulinum toxin (BOTOX®), which can exert a paralytic effect by binding to presynaptic cholinergic nerve terminals at the neuromuscular junction, is produced by the Gram-positive, rod-shaped, spore-forming, anaerobic bacterium Clostridium botulinum. It internalizes and inhibits the exocytosis of the neurotransmitter acetylcholine by decreasing the frequency of acetylcholine release

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and 65 years.
* Both sexes.
* Chronic migraine. Chronic migraine, defined as headaches on ≥15 days per month for ≥3 months, of which ≥8 days meet criteria for migraine without aura or respond to migraine-specific treatment according to International Classification of Headache Disorders-3 Beta.

Exclusion Criteria:

* Patients with medication over use headache.
* Bleeding disorders.
* Abnormal neurological examination.
* History of allergy to local anesthetics or BOTOX.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 12 weeks post-procedure
  The patients will be shown how to use the Visual Analogue Scale (VAS); 0-10 point where 0 = no pain and 10 = worst imaginable pain. VAS will be noted as well as after procedure, four-week, and 12-weeks period.

SECONDARY OUTCOMES:
Percentage of patients free of headache | 12 weeks post-procedure
  The percentage of patients free of headache at baseline (just before the procedure), after procedure, four-week, and 12-weeks period.
Headache relief rate | 12 weeks post-procedure
  Headache relief rate (percentage of patients with 50% or more reduction in headache intensity at four-week and 12-weeks period).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.